CLINICAL TRIAL: NCT00903682
Title: A Phase IIb, Multi-centre, Randomised, Double-blind, Active-controlled Trial Comparing the Neuropsychiatric Adverse Event Profile of Etravirine 400mg qd Versus Efavirenz 600mg qd in Combination With 2 Nucleoside/Nucleotide Reverse Transcriptase Inhibitors in ARV Therapy-naive HIV-1 Infected Subjects
Brief Title: A Clinical Trial Comparing the Tolerability of Etravirine to Efavirenz in Combination With 2 Nucleoside/Nucleotide Reverse Transcriptase Inhibitors in Treatment-naive HIV-1 Infected Patients
Acronym: SENSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR015751; TMC125VIR2038 (Other: Janssen-Cilag International NV); 2008-008655-42 (EudraCT Number)
Record Dates: First submitted 2009-05-14; First posted 2009-05-18 (Estimated); Results first posted 2011-03-07 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: HIV Infection; HIV; Acquired Immunodeficiency Syndrome
Keywords: HIV; Intelence; etravirine; ETR; TMC125; Sustiva; efavirenz; EFV; Non-nucleoside Reverse Transcriptase Inhibitor; NNRTI; treatment-naive
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — etravirine; efavirenz

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- etravirine (Experimental): etravirine (ETR TMC125) 400mg once daily (4x100mg tablet) + 2 NRTI + 1 EFV placebo tablet for 48 weeks
  Interventions: Drug: etravirine (ETR, TMC125)
- efavirenz (Active Comparator): efavirenz (EFV) 600mg once daily (1x600mg tablet) + 2 NRTIs + 4 ETR placebo tablets for 48 weeks
  Interventions: Drug: efavirenz (EFV)

INTERVENTIONS:
Drug: etravirine (ETR, TMC125) — 400mg once daily (4x100mg tablet) + 2 NRTI + 1 EFV placebo tablet for 48 weeks
  Arms: etravirine
Drug: efavirenz (EFV) — 600mg once daily (1x600mg tablet) + 2 NRTIs + 4 ETR placebo tablets for 48 weeks
  Arms: efavirenz

SUMMARY:
The purpose of this study is to compare the neuropsychiatric adverse event profiles of etravirine 400mg once daily versus efavirenz 600mg once daily, in combination with 2 N(t)RTIs, in approximately 150 treatment-naÃ-ve HIV-1 infected patients. Safety, tolerability and efficacy of both treatment arms will be assessed throughout the study.

DETAILED DESCRIPTION:
This is a phase IIb, randomised (study medication is assigned by chance), double-blind (neither the patient nor the study physician will know to which treatment group the patient is assigned) trial to assess the neuropsychiatric adverse event profile of etravirine (ETR) 400mg once daily versus efavirenz (EFV) 600mg once daily, each in combination with an investigator-selected background of 2 other anti-HIV drugs of the class nucleoside/nucleotide reverse transcriptase inhibitors (N[t]RTIs). The combination of N[t]RTIs to be chosen by the study physician can be abacavir (ABC)/lamivudine (3TC), zidovudine (AZT)/lamivudine (3TC) or tenofovir disoproxil fumarate (TDF)/emtricitabine (FTC). Approximately 150 Human Immuno-deficiency Virus type 1 (HIV-1) infected patients, who have never received any antiretroviral (ARV) treatment will be randomly assigned (like tossing a coin) to either the etravirine treatment group or the control group (efavirenz). The study period includes a screening period of maximum 6 weeks, a 48 week treatment period, an additional 2-8 weeks treatment until unblinding (study physician (and patient) will receive information to which treatment group the patient is assigned), followed by a 4 weeks follow-up period. The main purpose of this study is to gather further data on how many, how often, and how severe the central nervous system and psychiatric (neuropsychiatric) events are between the two treatment groups. In addition, the study will look at overall safety, tolerability and antiviral effectiveness between the two treatment groups. During the trial, patients' health will be monitored by physical examination, checking of vital signs (blood pressure / pulse), and laboratory testing on blood and urine samples. Also blood samples will be drawn to measure the antiviral effectiveness (i.e., decrease of the plasma viral load to a level <50 HIV-1 RNA (ribonucleic acid) copies/mL), immunology assessments (to assess the body's immune system) and pharmacokinetic (to measure the drug level in blood) analysis of etravirine. Patients will be asked to complete the "HIV Patient Symptoms Profile" (HIV PSP) Questionnaire at each visit, which contains questions relating to the impact on patients' current health and well-being. The study hypothesis is that the proportion of patients with at least one neuropsychiatric adverse event related to the study drug, observed between start of treatment (Baseline; BSL) through Week 12, is significantly lower in the etravirine group than in the efavirenz group. Patients will be taking blinded medication twice a day, administered orally (by mouth). Only one of the blinded doses will contain an active ingredient. Etravirine 400mg (or dummy-pills) - 4 tablets - should be taken once a day, following a meal, preferably breakfast. Efavirenz 600mg (or dummy-pill) - 1 tablet - should be administered once daily on an empty stomach, preferably at bedtime.The intake of the investigator-selected N[t]RTIs should be taken as instructed by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection
* In the judgement of the investigator, it is appropriate to initiate ARV therapy based on the patients medical condition and taking into account applicable guidelines for the treatment of HIV-1 infection
* Patient has access to an investigator-selected ARV regimen post-study in accordance with applicable guidelines for the treatment of HIV-1 infection
* HIV-1 plasma viral load at screening >= 5000 HIV-1 RNA (copies/ml)
* Predicted phenotypic sensitivity to the currently approved NNRTIs and to the N(t)RTIs in their background regimen at screening

Exclusion Criteria:

* Any previous treatment with a therapeutic HIV vaccine or use of ARVs, including use of NVP for the prevention of vertical HIV transmission
* The presence of at least one of the mutations that are specific indicators of transmitted (or primary) drug resistance
* Known infection with HIV-2 or with HIV-1 group O
* Category C AIDS defining illness, except stable Kaposi's Sarcoma, wasting syndrome if not progressive
* Pneumocystis jiroveci/carinii Pneumonia (PCP) that is considered not cured
* Specific grade 3 or 4 laboratory abnormalities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2009-06; Primary Completion 2010-02 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (33):
- Austria (2):
  - Salzburg
  - Vienna
- Denmark (2):
  - Aarhus
  - Odense
- France (5):
  - Bordeaux
  - Lyon
  - Nice
  - Paris
  - Strasbourg
- Germany (7):
  - Berlin
  - Bonn
  - Cologne
  - Essen
  - Frankfurt
  - Hamburg
  - Hanover
- Budapest, Hungary
- Israel (4):
  - Haifa
  - Jerusalem
  - Ramat Gan
  - Tel Aviv
- Romania (2):
  - Bucharest
  - Constanța
- Russia (2):
  - Moscow
  - Saint Petersburg
- Spain (4):
  - Barcelona
  - Granada
  - Madrid
  - Vigo
- Switzerland (2):
  - Bern
  - Zurich
- United Kingdom (2):
  - Brighton
  - London

REFERENCES:
- [Result] Nelson M, Stellbrink HJ, Podzamczer D, Banhegyi D, Gazzard B, Hill A, van Delft Y, Vingerhoets J, Stark T, Marks S. A comparison of neuropsychiatric adverse events during 12 weeks of treatment with etravirine and efavirenz in a treatment-naive, HIV-1-infected population. AIDS. 2011 Jan 28;25(3):335-40. doi: 10.1097/QAD.0b013e3283416873. PMID 21150563
- [Result] Gazzard B, Duvivier C, Zagler C, Castagna A, Hill A, van Delft Y, Marks S. Phase 2 double-blind, randomized trial of etravirine versus efavirenz in treatment-naive patients: 48-week results. AIDS. 2011 Nov 28;25(18):2249-58. doi: 10.1097/QAD.0b013e32834c4c06. PMID 21881478
- [Derived] Fatkenheuer G, Duvivier C, Rieger A, Durant J, Rey D, Schmidt W, Hill A, van Delft Y, Marks S; SENSE Study Team. Lipid profiles for etravirine versus efavirenz in treatment-naive patients in the randomized, double-blind SENSE trial. J Antimicrob Chemother. 2012 Mar;67(3):685-90. doi: 10.1093/jac/dkr533. Epub 2011 Dec 29. PMID 22210755

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Etravirine | Efavirenz
Started | 79 | 78
Completed | 63 | 63
Not Completed | 16 | 15
Not completed — Adverse Event | 6 | 13
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Pregnancy | 0 | 1
Not completed — Subject Reached A Virologic Endpoint | 1 | 1
Not completed — Subject Non-Compliant | 1 | 0
Not completed — Patient Couldn't Come For The Visit Due | 1 | 0
Not completed — For Resistent Profile (Excl Crit 2 Met) | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Etravirine: ETR 400mg once daily (4x100mg tablet) + 2 NRTIs + 1 EFV placebo tablet for 48 weeks
- Efavirenz: EFV 600mg once daily (1x600mg tablet) + 2 NRTIs + 4 ETR placebo tablets for 48 weeks
- Total: Total of all reporting groups
Arm/Group | Etravirine | Efavirenz | Total
Number analyzed (Participants) | 79 | 78 | 157
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 78 | 77 | 155
  >=65 years | 0 | 1 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 37.7 (9.52) | 37.6 (9.82) | 37.6 (9.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 18 | 30
  Male | 67 | 60 | 127
Region of Enrollment [Number; unit: participants]
  Austria | 3 | 4 | 7
  Denmark | 0 | 2 | 2
  France | 9 | 9 | 18
  Germany | 16 | 13 | 29
  Hungary | 5 | 3 | 8
  Israel | 4 | 5 | 9
  Italy | 9 | 6 | 15
  Romania | 6 | 10 | 16
  Russia | 9 | 8 | 17
  Spain | 12 | 9 | 21
  Switzerland | 1 | 3 | 4
  UK | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With at Least 1 Treatment-emergent Grade 1-4 Central Nervous System or Psychiatric Adverse Event
Description: Proportion of patients with at least 1 treatment-emergent Grade 1-4 Central Nervous System or psychiatric Adverse Event, observed between Baseline through Week 12 and judged by investigator to be at least possibly related to the study drug in ETR group versus EFV group. All Adverse Events were graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events ("DAIDS AE grading table"). Grade 1-4 covers all severities.
Time Frame: between baseline and 12 weeks
Population: The intent-to-treat (ITT) population has been defined as the set of all patients who were randomized and who have taken at least one dose of trial medication, regardless of their compliance with the protocol.
Measure: Number; unit: percentage of patients
Groups:
- Etravirine: Etravirine (ETR, TMC125) 400mg once daily (4x100mg tablet) + 2 non-nucleoside reverse transcriptase inhibitors (NRTIs) + 1 Efavirenz (EFV) placebo tablet for 48 weeks
Arm/Group | Etravirine | Efavirenz
Number analyzed (Participants) | 79 | 78
percentage of patients | 16.5 | 46.2
Statistical Analysis 1: Comparison: Etravirine vs Efavirenz; The hypothesis is that the proportion of patients with at least 1 treatment-emergent Grade 1-4 neuropsychiatric adverse event, observed between Baseline through Week 12 and judged to be at least possibly drug-related, is significantly lower in the ETR arm than in the EFV arm. Assuming a significance level of 5%, a sample size of 75 subjects per arm would provide over 90% power to detect a 29% difference in treatment-emergent, drug-related Grade 1-4 neuropsychiatric adverse events; Test type: Superiority or Other; p < 0.001, Regression, Logistic

2. Secondary Outcome: Antiviral Activity of ETR vs. EFV
Description: The proportion of patients with confirmed plasma viral load <50 copies/mL at Week 48 as assessed by Time to Loss of Virologic Response (TLOVR)
Time Frame: between baseline and week 48
Population: ITT: the set of all randomized patients who have taken at least 1 dose of trial medication, regardless of their compliance with the protocol.
Measure: Number; unit: Number of participants
Arm/Group | Etravirine | Efavirenz
Number analyzed (Participants) | 79 | 78
Number of participants | 60 | 58
Statistical Analysis 1: Comparison: Etravirine vs Efavirenz; Test type: Superiority or Other; Difference in proportion of response = 1.61, 95% CI 2-sided [-12.00 to 15.23] — Difference in proportion of response ETR minus EFV

3. Secondary Outcome: Antiviral Activity of ETR vs. EFV
Description: The proportion of patients with confirmed plasma viral load <200 copies/mL at Week 48 as assessed by Time to Loss of Virologic Response (TLOVR)
Time Frame: between baseline and week 48
Population: as for outcome 2
Measure: Number; unit: Number of participants
Arm/Group | Etravirine | Efavirenz
Number analyzed (Participants) | 79 | 78
Number of participants | 64 | 62

4. Secondary Outcome: Mean Change From Baseline in Neuropsychiatric and Total Tolerabililty Score
Description: The HIV Patient Symptoms Profile measures the tolerability of HIV treatment from the patient's perspective, using 14 concept scales in maximum 84 questions. The response options include a "no" or "yes" answer to "Did symptom occur?". If "yes", there is a problem scale which ranges from 1 = "I had this symptom and it was not a problem" to 5 = "I had this symptom and it was a severe problem". A neuropsychiatric tolerability score is composed as the sum of 21 items and ranges from 0 (best) to 105 (worse). A total Tolerability score (ie, the sum of all items) ranges from 0 (best) to 420 (worse)
Time Frame: between baseline and week 48
Population: as for outcome 2
Measure: Mean (Standard Error); unit: points on a scale
Arm/Group | Etravirine | Efavirenz
Number analyzed (Participants) | 75 | 74
points on a scale
  Total Tolerability Score | -0.04 (0.03) | -0.01 (0.04)
  Neuropsychiatric Tolerability Score | -0.04 (0.06) | -0.07 (0.07)

5. Secondary Outcome: Neuropsychiatric Adverse Events by Week 48
Description: The percentage of patients with at least 1 treatment emergent Grade 1 -4 neurologic or psychiatric adverse event, judged by the investigator to be at least possibly related to the study drug.
Time Frame: from baseline to week 48
Population: as for outcome 2
Measure: Number; unit: percentage of patients
Arm/Group | Etravirine | Efavirenz
Number analyzed (Participants) | 79 | 78
percentage of patients | 20.3 | 52.6

6. Secondary Outcome: Mean Change From Baseline in CD4+ Cell Count
Description: The mean change in CD4+ cell count from baseline was calculated with a last observation carried forward method; i.e. the last observed value was carried forward, irrespective of the reason for discontinuation.
Time Frame: at baseline and week 2, 6, 12, 24, 36 and 48
Population: as for outcome 2
Measure: Mean (Standard Error); unit: number of cells/L (x10^6)
Arm/Group | Etravirine | Efavirenz
Number analyzed (Participants) | 74 | 74
number of cells/L (x10^6)
  Week 2 | 69.96 (9.82) | 72.45 (11.33)
  Week 6 | 128.14 (13.19) | 121.62 (13.96)
  Week 12 | 143.24 (13.56) | 151.46 (16.68)
  Week 24 | 182.01 (16.48) | 174.08 (14.85)
  Week 36 | 213.45 (19.11) | 180.18 (15.12)
  Week 48 | 205.11 (20.07) | 221.39 (18.31)

7. Secondary Outcome: Resistance Determinations
Description: The evolution of viral genotype and phenotype was assessed by the number of patients with resistance-associated mutations emerging at the endpoint. A mutation was considered emerging if it was present at endpoint and not present at baseline or any pre-baseline assessment. (NNRTI = non-nucleoside reverse transcriptase inhibitor; NRTI = nucleoside reverse transcriptase inhibitor; RAM = resistance-associated mutation, IAS-USA = International AIDS Society - USA)
Time Frame: at baseline and all subsequent visits until week 48 in case if virologic failure
Population: as for outcome 2
Measure: Number; unit: number of participants
Arm/Group | Etravirine | Efavirenz
Number analyzed (Participants) | 79 | 78
number of participants
  >= 1 successful genotype after baseline | 11 | 9
  >= 1 IAS-USA NRTI RAMs | 0 | 2
  >= 1 NRTI Surveillance Drug Resistance Mutation | 0 | 2
  >= 1 NNRTI RAMs | 2 | 3
  no NRTI or NNRTI RAMs | 9 | 6

ADVERSE EVENTS:
Time Frame: Adverse events represented here were collected between signing of informed consent and the visit at week 48.
Arm/Group | Etravirine | Efavirenz
Serious Adverse Events (participants affected / at risk) | 11/79 | 6/78
Other Adverse Events (participants affected / at risk) | 54/79 | 62/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etravirine (N=79) | Efavirenz (N=78)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pulmonary Tuberculosis (Infections and infestations) | 0 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Anal Fissure (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Anal Abscess (Infections and infestations) | 0 | 1
Anogenital Warts (Infections and infestations) | 1 | 0
Secondary Syphilis (Infections and infestations) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 1
Joint Ankylosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Benign Ovarian Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Urethral Stenosis (Renal and urinary disorders) | 1 | 0
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Abortion Induced (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etravirine (N=79) | Efavirenz (N=78)
Vertigo (Ear and labyrinth disorders) | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 8 | 9
Nausea (Gastrointestinal disorders) | 7 | 13
Vomiting (Gastrointestinal disorders) | 2 | 6
Asthenia (General disorders) | 3 | 5
Pyrexia (General disorders) | 5 | 5
Influenza (Infections and infestations) | 6 | 1
Nasopharyngitis (Infections and infestations) | 17 | 6
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 7
Dizziness (Nervous system disorders) | 3 | 17
Headache (Nervous system disorders) | 13 | 11
Somnolence (Nervous system disorders) | 2 | 5
Abnormal Dreams (Psychiatric disorders) | 2 | 9
Insomnia (Psychiatric disorders) | 2 | 8
Nightmare (Psychiatric disorders) | 3 | 7
Sleep Disorder (Psychiatric disorders) | 4 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 7
Anaemia (Blood and lymphatic system disorders) | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 6 | 3
Fatigue (General disorders) | 5 | 6
Bronchitis (Infections and infestations) | 5 | 5
Pharyngitis (Infections and infestations) | 4 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 7 | 3
Disturbance in Attention (Nervous system disorders) | 1 | 4
Anxiety (Psychiatric disorders) | 1 | 4
Depression (Psychiatric disorders) | 1 | 5
Rash (Skin and subcutaneous tissue disorders) | 5 | 2
Hot Flush (Vascular disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the Sponsor for review at least 60 days prior to submission for publication or presentation. No paper that incorporates Confidential Information will be submitted for publication without Sponsor's prior written consent. If requested in writing, such publication will be withheld for up to an additional 60 calendar days. A publication from the individual Study site data will not be published until the combined results have been published.